CLINICAL TRIAL: NCT01675219
Title: Treatment of Ta Bladder Cancer in High Risk of Recurrence - Fluorescence Cystoscopy With Optimized Adjuvant Mitomycin-C (FinnBladder 9)
Brief Title: Fluorescence Cystoscopy and Optimized MMC in Recurrent Bladder Cancer (FinnBladder 9)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Finnbladder (Other)
Responsible Party: Principal Investigator, Peter Boström, MD, PhD, Turku University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FinnBladder 9; 2012-000559-15 (EudraCT Number)
Record Dates: First submitted 2012-08-25; First posted 2012-08-29 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; recurrence; photodynamic diagnosis; PDD; cost analysis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group B (Experimental): Blue light TUR-BT with no adjuvant instillations
  Interventions: Procedure: blue light TUR-BT; Drug: single immediate chemotherapy instillation
- Group A (Active Comparator): White light TUR-BT with no adjuvant instillations
  Interventions: Procedure: white light TUR-BT; Drug: single immediate chemotherapy instillation
- Group C (Experimental): White light TUR-BT with six weekly optimized mitomycin-C instillations.
  Interventions: Drug: optimized MMC; Drug: single immediate chemotherapy instillation
- Group D (Experimental): Blue light (PDD) TUR-BT with six weekly optimized mitomycin-C instillations.
  Interventions: Procedure: blue light TUR-BT; Drug: optimized MMC; Drug: single immediate chemotherapy instillation

INTERVENTIONS:
Procedure: white light TUR-BT — traditional transurethral bladder tumor resection
  Arms: Group A
Procedure: blue light TUR-BT — photodynamic transurethral bladder tumor resection
  Arms: Group B; Group D
Drug: optimized MMC — six weekly optimized mitomycin-C instillations
  Other Names: optimized mitomycin-C
  Arms: Group C; Group D
Drug: single immediate chemotherapy instillation — single immediate post TUR-BT epirubicin (2mg/ml, total of 100 ml) instillation
  Other Names: single instillation

SUMMARY:
Bladder cancer (BC), the second most common urological malignancy, is an important public health issue. One of the main challenges in the treatment of bladder cancer if the prevention of recurrences of non-invasive tumors, which is also associated with significant costs.

The current study will investigate optimal treatment of patients with bladder cancer with high risk of tumor recurrence but low risk of progression. The main interest is comparison of photodynamic (PDD) bladder tumor resection (TUR-BR)to traditional TUR-BT. Also the efficacy of adjuvant optimized mitomycin-C is compared to patients with no adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

- Primary papillary bladder cancer at high risk for further recurrence as defined as follows:

Number of primary tumors ≥2, OR Size of solitary primary tumor ≥ 3 cm, OR Recurrent papillary tumors

* Histologically proven Ta bladder cancer
* Histological grade 1-2 (WHO 1973 grading system) or papillary urothelial neoplasm of low malignant potential (PUNLMP) or low grade (WHO 2004 grading system) bladder cancer
* Written informed consent is required from every eligible patient

Exclusion Criteria:

* Grade 3 tumors (WHO 1973 grading system), or high grade tumors (WHO 2004 grading system)
* CIS (carcinoma in situ)
* Suspicion or evidence of papillary tumors or CIS of the upper urinary tract
* Non-TCC (transitional cell carcinoma, i.e. urothelial carcinoma) bladder cancer
* Suspicion or previous history of the patient not tolerating intravesical instillations
* Known allergy to MMC or hexaminolevulinate (HAL, Hexvix®)
* Urethral stricture, stone disease, chronic urinary tract infection or any other urological condition that may compromise study participation (as judged by treating physician)
* Pregnancy or lactating patient
* Other non-cured malignancy (excepting skin basalioma or cancer in situ of the cervix uteri or any other malignancy in remission ≥5 years)
* Age < 18 years
* Expected survival time less than one year
* Expected poor compliance (e.g. some severe psychiatric disorders, antisocial behaviour, or dementia)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-12; Primary Completion 2021-12 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
bladder cancer recurrence rate | 2 years
  any bladder cancer recurrence at 2 years.

SECONDARY OUTCOMES:
Bladder cancer progression | 2 years
  bladder cancer progression to T2 or higher
Treatment failure | 2 years
  progression, recurrence or side effects preventing completing the trial
mortality | 2 years
  death due bladder cancer or other reasons

OTHER OUTCOMES:
costs | 2 years
  For analysis of cost-effectiveness. All bladder cancer treatment and treatment complications related costs are included.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Boström, MD, PhD, Principal Investigator — Turku University Hospital; Eero Kaasinen, Md, PhD, Study Director — Hyvinkää District Hospital
Locations (10):
- Finland (10):
  - HYKS Peijas Hospital, Helsinki
  - Hyvinkää District Hospital, Hyvinkää
  - Kuopio University Hospital, Kuopio
  - Mikkeli Central Hospital, Mikkeli
  - Oulu University Hospital, Oulu
  - Satakunnan keskussairaala, Pori
  - Seinäjoki Central Hospital, Seinäjoki
  - Hatanpään sairaala, Tampere
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Sell V, Ettala O, Perez IM, Jarvinen R, Pekkarinen T, Vaarala M, Seppanen M, Liukkonen T, Marttila T, Aaltomaa S, Bostrom PJ. Awareness of Smoking as a Risk Factor in Bladder Cancer: Results from the Prospective FinnBladder 9 Trial. Eur Urol Focus. 2022 Sep;8(5):1246-1252. doi: 10.1016/j.euf.2022.01.012. Epub 2022 Jan 31. PMID 35094962